CLINICAL TRIAL: NCT06239389
Title: Comparison Of Efficacy And Safety Of Thalidomide Vs Hydroxyurea In Thalassemia Patients: A Single-Centre Pilot Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIBD/IRB-236/21-2021.
Record Dates: First submitted 2023-12-23; First posted 2024-02-02 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Beta-Thalassemia
Keywords: thalidomide,; hydroxyurea; hemoglobin F inducers; beta thalassemia
MeSH Terms: conditions — beta-Thalassemia | interventions — Thalidomide; Hydroxyurea

STUDY DESIGN:
Intervention Model Description: Patients were divided into 2 groups, one received hydroxyurea second group received thalidomide.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hydroxyurea (Active Comparator): Hydroxyurea is available in oral dosage form which is capsule. frequency: once a day duration: at every 24 hours dose: 15/mg/kg/day.
  Interventions: Drug: Thalidomide 100mg
- Thalidomide (Experimental): Thalidomide is available in oral dosage form which is capsule. frequency: once a day at night duration: at every 24 hours dose:50 mg / day (in patients >10-13 years) while the adult dose was 100 mg /day (age >13 Years)
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Thalidomide 100mg — Thalidomide is available in capsulated form in the strength of 100 mg and 50 mg. It was given according to the weight of the patient. Due to somnolence, it was advised to give at night only.
  Other Names: thalido
  Arms: hydroxyurea
Drug: Hydroxyurea — Hydroxyurea is available in capsulated form under the brand of hydrea. Its available strength is 500 mg . Dosing depends upon weight of patient, that is 15mg/kg/day. so patients unable to take full capsule due to low weight, was advised to take hydroxyurea syrup.
  Other Names: Hydrea
  Arms: Thalidomide

SUMMARY:
The goal of this study is to compare the effectiveness and safety of two hemoglobin F inducer. This is single centered interventional pilot study is to compare the efficacy and safety parameters in beta thalassemia patients. As this is a pilot study, the investigator took a small number of patients. The Sample size was calculated by the World health organization sample size calculator. After screening 39 patients and 24 patients were eligible for enrollment in this study.

The main objective was to evaluate safety of both drugs in genetic disorder like thalassemia. for safety evaluation, hematological parameters were evaluated that includes total bilirubin , indirect bilirubin, Serum Glutamate Pyruvate Transaminase, serum glutamic-oxaloacetic transaminase, urea, creatinine and lactate dehydrogenase were monitored . Moreover to evaluate the efficacy of drug, hematological parameters that includes hemoglobin, red blood cells , nucleated red blood cells , reticulocytes count, Red blood cells indices ( mean corpuscular hemoglobin, mean corpuscular volume and mean corpuscular hemoglobin concentration) , white blood cells and platelets were done. Another important parameters to evaluate the efficacy of hemoglobin F inducer is transfusion frequency.

Test were done at baseline and after completion of study means after 06 months.

ELIGIBILITY:
Inclusion Criteria:

* Know case of beta thalassemia age between 10-30 years

Exclusion Criteria:

* Patients on any other haemoglobin F inducer or erythropoietin.
* Patients with co-morbidities like cardiopulmonary and neurological disease
* Pregnant, lactating women.
* Patient did not willing to take contraceptive measures.
* Participants with history of thrombosis.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
comparison of hemoglobin | 06 months
  Hemoglobin
comparison of red blood cells | 06 months
  Red blood cells
comparison of Mean corpuscular volume | 06 months
  Mean corpuscular volume
comparison of Mean Corpuscular Hemoglobin | 06 months
  Mean Corpuscular Hemoglobin
comparison of Mean Corpuscular Hemoglobin concentration | 06 months
  Mean Corpuscular Hemoglobin concentration
comparison of Indirect bilirubin | 06 months
  Indirect bilirubin
comparison of Total Bilirubin | 06 months
  Total Bilirubin
comparison of Serum glutamic pyruvic transaminase | 06 months
  Serum glutamic pyruvic transaminase
comparison of glutamic-oxaloacetic transaminase | 06 months
  glutamic-oxaloacetic transaminase
comparison of white blood cells | 06 months
  white blood cells
comparison of platelets | 06 months
  Platelets
comparison of urea | 06 months
  Urea
comparison of creatinine | 06 months
  Creatinine
comparison of Lactate dehydrogenase baseline and after the completion of study. | 06 months
  Lactate dehydrogenase
comparison of tranfusion frequency baseline and after the completion of study. | 06 months
  Transfusion interval

CONTACTS AND LOCATIONS:
Overall Officials: Safia Mehmood khan, MPHIL, Principal Investigator — National institute if blood diseases and bone marrow transplantation
Locations (1):
- National Institute of Blood Diseases and Bone Marrow Transplantation, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No